CLINICAL TRIAL: NCT00969657
Title: Prospective Validation of a Predictive Model for Pathologic Complete Response After Chemoradiotherapy in Rectal Cancer: A Prognostic Study
Brief Title: Validation of a Predictive Model After Complete Response in Rectal Cancer
Acronym: Thunder
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 6050; 09-03-023
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer stage I-III; concurrent chemoradiotherapie; response prediction
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum,plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background of the study:

Prediction of rectal tumor response after chemoradiotherapy (CRT) might be helpful in individualizing treatment strategies, i.e., selecting patients who need less invasive surgery or another radiotherapy strategy instead of resection. For rectal cancer it is known that 10-30% of the patients will respond with a pathologic complete response (pCR) after CRT. From a retrospective study with multivariate analysis of both clinical and 2-[18F] fluoro-2-deoxy-D-glucose and positron emission tomography (FDG-PET) data, it was found that adding FDG-PET data collected before and after CRT leads to a more predictive model compared to evaluating only pretreatment clinical data. To validate this model, this registration study is proposed. Furthermore, it has been found that FDG-PET during treatment is very predictive for response and a more favorable time point to adapt treatment. Also, there are indications that adding blood biomarkers to the data, results in higher accuracy for response prediction compared to clinical and imaging data alone. Therefore, FDG-PET during treatment and blood sampling are included in the protocol to improve the accuracy of the prediction models.

Objective of the study:

The long-term research objective is to be able to select rectum cancer patients who could receive a less invasive treatment. If prediction of response is possible, surgery may be avoided when complete response after chemoradiotherapy is expected or performed with smaller incisions if stage reduction is significant. This support decision system helps to individualize patient treatment and can improve the quality of life for the patient.

Study design:

28x radiotherapy. On day 15 of radiotherapy en 8 weeks after radiotherapy: 1 PET-CT scan Before radiotherapy, on day 15 and 8 weeks after radiotherapy: blood sample taken.

DETAILED DESCRIPTION:
General objective

The long-term research objective is to be able to select rectum cancer patients who could receive a less invasive treatment. If prediction of response is possible, surgery may be avoided when complete response after chemoradiotherapy is expected or performed with smaller incisions if stage reduction is significant. This support decision system helps to individualize patient treatment and can improve the quality of life for the patient.

Aim of the study

The main aim is to validate a predictive model for pathologic complete response (ypT0N0) in rectal cancer patients treated with chemoradiotherapy by multi-centric prospective data collection. The second aim is to collect extra data for improvement of the accuracy of the prediction models with new variables. This new model will be validated later in the model development process.

Hypothesis

General hypothesis:

The validated accuracy of predictive models for pathologic complete response after chemoradiotherapy in rectal cancer patients is high enough to tailor treatment (surgery/non-surgery and/or administer extra radiation boosts) in clinical practice.

Specific hypotheses:

1. The performance of the developed models on the validation data is at least equal to the performance achieved during the model development process.
2. The performance of a new model based on the addition of variables performs better than the previous model

ELIGIBILITY:
Inclusion Criteria:

* Histological proven rectal cancer
* UICC stage I-III
* Only primary tumors; no recurrences
* Only concurrent chemoradiotherapy treatment
* Willing and able to comply with the study prescriptions
* 18 years or older
* Have given written informed consent before patient registration
* No previous radiotherapy to the pelvis

Exclusion Criteria:

* No adenocarcinoma histology
* History of prior pelvis radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (ypT0N0) | 8-12 weeks after long-series chemoradiotherapy

SECONDARY OUTCOMES:
Several extra outcomes are registered for research: Local relapse at 2 years, metastases free survival, survival and relapse free survival | five years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, prof, Study Director — Maastricht Radiation Oncology
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Roelofs E, Dekker A, Meldolesi E, van Stiphout RGPM, Valentini V, Lambin P. International data-sharing for radiotherapy research: an open-source based infrastructure for multicentric clinical data mining. Radiother Oncol. 2014 Feb;110(2):370-374. doi: 10.1016/j.radonc.2013.11.001. Epub 2013 Dec 3. PMID 24309199